CLINICAL TRIAL: NCT00057460
Title: Effects of AMPA Receptor Blockade on Human Cortical Excitability - A Pilot Study
Brief Title: Effect of Talampanel (an AMPA Receptor Blocker) on Brain Activity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030147; 03-N-0147
Record Dates: First submitted 2003-04-02; First posted 2003-04-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-05

CONDITIONS: Healthy
Keywords: Antiepileptic Drug; Neuroprotection; Seizure Disorder; TMS Stimulation; EEG; AMPA Antagonist; Dosing; Transcranial Magnetic Stimulation; Healthy Volunteer; HV
MeSH Terms: conditions — Epilepsy | interventions — talampanel

INTERVENTIONS:
Drug: Talampanel

SUMMARY:
This study will use transcranial magnetic stimulation (TMS) and electroencephalography (EEG) to test the safety of an experimental anti-epileptic drug called Talampanel and learn how it affects brain activity. Talampanel blocks a type of brain receptor called AMPA; inhibiting this receptor may result in anti-seizure activity.

TMS stimulates the outer part of the brain, called the cortex. For this procedure, an insulated wire coil is placed on the subject's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. This may cause a pulling sensation on the skin under the coil and muscle twitching in the face, arm, or leg.

EEG records the electrical activity of the brain, in the form of brain waves. For this procedure, electrodes (metal discs with a conductive gel) attached to wires are affixed to the scalp with a paste and the brain activity is recorded.

Healthy normal volunteers between 18 and 45 years of age may participate in this study. Candidates will be screened with a physical and neurological examination, electrocardiogram (EKG), blood tests, and blood pressure measurement. Women who are pregnant or nursing are excluded from the study.

Participants will come to the NIH Clinical Center for three testing sessions, at least 1 week apart, and a final follow-up visit. The procedure for each test session is as follows:

7 AM - Blood pressure is measured, EKG and EEC leads are placed, a heparin lock is inserted, and a blood sample is drawn. The heparin lock is a thin needle enclosed in a thin plastic tube. The needle guides the tube into a vein and is then removed, leaving the tube in place. The indwelling tube allows multiple blood samples to be drawn without repeated needle sticks.

8 - 9 AM - TMS followed by EEG recording.

9 AM - Administration of Talampanel or placebo (pill with no active ingredient) by mouth.

10 AM - Blood sample #2.

10 AM -11 AM - TMS, followed by EEG recording every 5 minutes.

11 AM - Blood sample #3.

12 PM - Blood sample #4.

11 AM - 1 PM - EEG recording every 5 minutes/

4 PM - Blood sample #5.

5 PM - Discharge from Clinical Center.

At the final follow-up visit, the participant will talk with the doctor and have one final blood draw.

DETAILED DESCRIPTION:
Objectives. The purpose of this pilot study is to identify human neurophysiological parameters that are sensitive to talampanel, as assessed by transcranial magnetic stimulation (TMS) and electroencephalography (EEG). Talampanel is a highly selective, orally active antagonist of the AMPA (alpha-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid) receptor. The study will test two hypotheses: (1) talampanel will, in a dose-dependent fashion, suppress the motor-evoked potential (MEP) amplitude and intracortical facilitation as determined by TMS, and (2) talampanel will, in a dose-dependent fashion, cause alterations in EEG power within specific frequency bands. We plan to administer a low (25 mg) and high (50 mg) dose of talampanel and placebo to normal volunteers and measure various TMS and EEG parameters that we hypothesize may be influenced by AMPA receptor blockade. We will simultaneously assay serum levels of talampanel. We will use statistical tests to correlate changes in the TMS and EEG measures with drug concentration. The results of this study will allow us to undertake a follow-up study in which we will determine the effects of AMPA receptor blockade by talampanel on human motor and cognitive function. Our ultimate goal is to determine whether drug-induced blockade of AMPA receptors can be achieved without unacceptable neurological impairment.

Study population. This will be a blinded and placebo-controlled pilot study using 12 normal volunteers.

Design. Normal volunteers accepted into the study will be subjected to the following exams: (a) TMS determination of MEP amplitude and paired-pulse testing at baseline and at peak serum levels after drug or placebo administration, (b) digital EEG recording for 1 h at baseline before administration of drug or placebo and during a period of 3 h after administration. Samples for serum chemistry, liver function tests, hematology, and urinalysis will be obtained at admission, at discharge, and in every clinic visit during the study. Blood samples for determining serum talampanel levels will be obtained at 1, 2, 3, and 8 h after drug administration. MEPs at interstimulus intervals of 2 to 20 ms will be compared among subjects before and after drug administration, by a repeated measures analysis of variance. Talampanel levels will be correlated with MEP amplitudes by regression analysis.

Clinical endpoint. This pilot study will identify information on the best TMS interstimulus interval or intervals for measuring changes in cortical excitability after AMPA blockade, as well as the EEG frequency band most sensitive to AMPA blockade with talampanel. Because talampanel is a highly selective AMPA receptor antagonist, we will be able to infer that the parameters that are sensitive to talampanel can be used as empirical assays of AMPA receptor function in humans.

ELIGIBILITY:
INCLUSION CRITERIA:

Study subjects must be 18-45 years old (inclusive).

Study subjects must give informed consent in writing prior to entering the study.

Study subjects must be able to participate for the full term of the trial.

EXCLUSION CRITERIA:

Any of the following conditions is cause for exclusion from the study:

Any illness requiring chronic drug therapy with one of the following drugs: Depakote (valproic acid), Hismanal (astemizole), Propulsid (cisapride), Allegra (fexofenadine), Seldane (terfenadine), Luvox (fluvoxamine), Felbamate (felbatol), Tiagabine (vigabatrin), hepatic enzyme inducers such as Tagamet (cimetidine), and -azole antifungals such as Flagyl (metronidazole), Diflucan (fluconazole), and Nizoral (ketoconazole).

History of a psychiatric disorder, under the care of a psychiatrist, or on medications for treatment of a psychiatric disorder.

Known sensitivity or allergy to talampanel or related compounds.

Use of illicit drugs, binge drinking, or alcoholism as per medical history inventory.

Exposure to any other investigational drug within 12 weeks prior to randomization.

Magnetic stimulation will not be performed in people who have pacemakers, implanted pumps or stimulators, or who have metal objects inside the eye or skull.

Being under the age of 18 years or over the age of 45 years.

Pregnant or lactating.

Cardiac, pulmonary, or neurological problems as determined by medical history, EKG, and examination by a physician.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2003-04; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Anand S, Hotson J. Transcranial magnetic stimulation: neurophysiological applications and safety. Brain Cogn. 2002 Dec;50(3):366-86. doi: 10.1016/s0278-2626(02)00512-2. PMID 12480484
- [Background] Belayev L, Alonso OF, Liu Y, Chappell AS, Zhao W, Ginsberg MD, Busto R. Talampanel, a novel noncompetitive AMPA antagonist, is neuroprotective after traumatic brain injury in rats. J Neurotrauma. 2001 Oct;18(10):1031-8. doi: 10.1089/08977150152693728. PMID 11686490
- [Background] Berardelli A, Rothwell JC, Thompson PD, Hallett M. Pathophysiology of bradykinesia in Parkinson's disease. Brain. 2001 Nov;124(Pt 11):2131-46. doi: 10.1093/brain/124.11.2131. PMID 11673316